CLINICAL TRIAL: NCT04920539
Title: In Vivo Study of THC-induced Immune-genome Changes at Single Cell Solution in HIV-infected Humans
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000030067; R01DA052846 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-06-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Healthy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Delta-9-THC (Experimental): Active Delta-9-THC (0.03 mg/kg) administered intravenously.
  Interventions: Drug: Active Delta-9-THC

INTERVENTIONS:
Drug: Active Delta-9-THC — Active Delta-9-THC (0.03 mg/kg) administered intravenously.

SUMMARY:
In this study, the investigators hypothesize that THC alters the immunogenome in a cell type-specific fashion and alters cytokine production via epigenetic regulatory mechanisms and that these alterations differ between HIV-infected and HIV-uninfected host genomes.

DETAILED DESCRIPTION:
In this study, the investigators hypothesize that THC alters the immunogenome in a cell type-specific fashion and alters cytokine production via epigenetic regulatory mechanisms and that these alterations differ between HIV-infected and HIV-uninfected host genomes. To test these hypotheses, the investigators propose defining the epigenomic and transcriptomic alterations at single cell resolution in peripheral blood mononuclear cells by administering THC to humans with and without HIV infection. The THC-associated epigenomic/transcriptomic alterations will be linked to genomic variants to understand the causal effects of THC response in immune cells.

ELIGIBILITY:
Inclusion Criteria (HIV-infected group):

* HIV-positive
* Good medication adherence
* Negative urine toxicology for drugs of abuse (including cannabis)
* Good mental and physical health (other than HIV) as determined by history, psychiatric interview, collateral information, physical and laboratory examinations, ECG, and vital signs.

Inclusion Criteria (HIV-uninfected group):

* HIV-negative
* Negative urine toxicology for drugs of abuse (including cannabis)
* Good mental and physical health as determined by history, psychiatric interview, collateral information, physical and laboratory examinations, ECG, and vital signs.

Exclusion Criteria (common to both groups):

* Major medical conditions, e.g., myocardial infarction, hypertension, etc.
* Positive pregnancy test and lactation;
* Weight greater than 166 kg (365 lbs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Gene Expression Alteration | Blood samples will be collected to measure changes in gene expression altered by THC before study drug infusion and at 70, 140, and 300 minutes after study drug infusion.
  Quantity of each gene is measured via sequence transcriptome, and significant differences of quantified gene pre- and post-THC infusion will be identified as THC-induced gene expression alteration.
Change in Cytokine Profile | Blood samples will be collected to measure changes in cytokine profile before study drug infusion and at 70, 140, and 300 minutes after study drug infusion.
  Cytokine profile will be measured using Luminex Performance Human Cytokine Discovery panel before and after study drug infusion. The 45 cytokines selected based on their established role in immune functioning are: CCL2/MCP-1, CCL3/MIP-1a, CCL4/MIP-1b, CCL5/RANTES, CCL11/Eotaxin, CCL19/MIP-3b, CCL20/MIP-3a, TNFSF5, CX3CL1/Fractalkine, CXCL1/GROa, CXCL2/GROb, CXCL10/IP-10, EGF, FGF2, FLT3L, G-CSF, GM-CSF, Granzyme B, IFN-a2, IFN-b, IFN-g, IL-1a, IL-1b, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8/CXCL8, IL-10, IL-12 p70, IL-13, IL-15, IL-17A, IL-17E, IL-33, PD-L1, PDGF-AA, PDGF-AB/BB, TGF-a, TNF-a, TNFSF10, VEGF.
Change in Gene Expression Alteration by THC between HIV-positive and HIV-negative Groups | Blood samples will be collected to measure change in gene expression altered by THC before study drug infusion and at 70, 140, and 300 minutes after study drug infusion.
  Quantity of each gene is measured via sequence transcriptome, and significant differences of quantified gene pre- and post-THC infusion are identified as THC-induced gene expression alteration. Results will be compared between HIV-positive and HIV-negative subjects.
Change in Cytokine Profile by THC between HIV-positive and HIV-negative Groups | Blood samples will be collected to measure changes in cytokine profile by THC before study drug infusion and at 70, 140, and 300 minutes after study drug infusion.
  Cytokine profile will be measured using Luminex Performance Human Cytokine Discovery panel before and after study drug infusion. Results will be compared between HIV-positive and HIV-negative subjects. The 45 cytokines selected based on their established role in immune functioning are: CCL2/MCP-1, CCL3/MIP-1a, CCL4/MIP-1b, CCL5/RANTES, CCL11/Eotaxin, CCL19/MIP-3b, CCL20/MIP-3a, TNFSF5, CX3CL1/Fractalkine, CXCL1/GROa, CXCL2/GROb, CXCL10/IP-10, EGF, FGF2, FLT3L, G-CSF, GM-CSF, Granzyme B, IFN-a2, IFN-b, IFN-g, IL-1a, IL-1b, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8/CXCL8, IL-10, IL-12 p70, IL-13, IL-15, IL-17A, IL-17E, IL-33, PD-L1, PDGF-AA, PDGF-AB/BB, TGF-a, TNF-a, TNFSF10, VEGF.

SECONDARY OUTCOMES:
Perceptual Alterations | Perceptual alterations will be measured before study drug infusion and 70, 140, and 300 minutes after study drug infusion.
  Perceptual alterations will be measured using scales such as the Clinician Administered Dissociative Symptoms Scale (CADSS), a scale consisting of 19 self-report items and 8 clinician-rated items (0 = not at all, 4 = extremely) that we have shown to be sensitive to THC effects. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Cannabis Subjective Effects | Cannabis subjective effects will be measured before study drug infusion and 70, 140, and 300 minutes after study drug infusion.
  Various feeling states associated with cannabis intoxication will be measured using a self-reported visual analog scale of feeling states ("high", "calm and relaxed", and "tired") associated with cannabis effects. Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 100 mm line (0 = not at all, 100 = extremely). These data will be captured to validate that the experiment is relevant to cannabis effects.
Cannabinoid Relevant Molecules | Blood will be collected before study drug infusion and at 70, 140, and 300 minutes after study drug infusion.
  Blood will be sampled for cannabinoid relevant molecules before and after study drug infusion. Cannabinoid relevant molecules will include THC and THC-COOH levels.
Change in total immediate recall on the RAVLT. | The RAVLT will be administered prior to study drug administration at approximately 25 minutes after study drug administration.
  Memory, attention, and executive function will be measured before and after study drug administration using the Rey Auditory Verbal Learning Task (RAVLT).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University Professor of Psychiatry
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States